CLINICAL TRIAL: NCT03495219
Title: Subjects Ability to Control Pressure in the Lower Esophageal High Pressure Znoe (HPZ) During Manometry.
Brief Title: Can Individuals Control Pressure in Their Esophagus.
Acronym: manometry
Status: Withdrawn | Type: Observational
Why Stopped: Unable to use manometry lab.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, C. Joseph Yelvington P.T., D.P.T., Principal Investigator, Mayo Clinic
Other Study IDs: 17-003796
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Esophageal Manometry: Esophageal manometry is a test to assess motor function of the upper esophageal sphincter, esophageal body and lower esophageal sphincter
  Interventions: Procedure: Esophageal Manometry

INTERVENTIONS:
Procedure: Esophageal Manometry — A catheter inserted through the nares, post appropriate anesthetization. The subject is then given 8 - 10 sips of water or semi viscous fluid during the routine study. At the conclusion of the clinical portion of the examination the manometer catheter is typically removed by the technician at that point. For the purposes of this research study the catheter will remain in place to examine pressures specifically at the lower end of the esophagus during various breathing patterns and training activities to see if pressures can be increased with instruction.

SUMMARY:
To establish to what degree individuals can increase esophageal high pressure zone (HPZ) after instruction in deep breathing as evidenced by concurrent manometric pressure readings.

DETAILED DESCRIPTION:
Pressure in the lower esophagus has been negatively associated with reflux symptoms: the lower the pressure, the more reflux symptoms. This pressure can be augmented with deep abdominal breathing. This can be detected during esophageal manometry, when a pressure catheter is placed into the esophagus. Manometry is routinely done for swallowing disorders.

This study will take place just after a routine manometry test, when the subject still has the catheter in place. All that is required for the research portion is to observe manometry readings while they breathe, then when they deep breath, then breathe after they have been cued or coached to deep abdominal breathing. This is done in sequence to establish how quickly this pressure can be improved.

This coached breathing is then prescribed as a routine exercise and long term follow up performed via phone to see how their reflux symptoms have responded.

ELIGIBILITY:
Inclusion Criteria:

-Eligibility is forwarded to all individuals undergoing routine esophageal manometry. They would have had to have met all eligibility criteria for this procedure.

Exclusion criteria:

-Individuals undergoing modified barium swallow studies (MBSS). Exclusion from MBSS would preclude inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults undergoing outpatient ambulatory procedures at Mayo Clinic Jacksonville.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-01-02 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Reflux Symptom Index Score (RSI) | 3 months.
  Does intervention reduce RSI score from before intervention to follow up.

SECONDARY OUTCOMES:
Association of RSI to resting manometry pressure in the lower esophagus | 1 day
  At rest, is basal esophageal pressure associated with subjects RSI scores?
Can lower esophageal pressure can be increased by instruction/coaching by a physical therapist. | 1 day
  Verbal, tactile coaching on diaphragm recruitment will be given while under manometry to establish the ability of subjects to improve lower esophageal pressure.

CONTACTS AND LOCATIONS:
Overall Officials: C J Yelvington, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: Undecided
What may be released include: study protocol, statistical analysis, clinical study report. Should this want to be replicated at other Mayo sites.

REFERENCES:
- [Background] Sun XH, Ke MY, Wang ZF, Fang XC. [Roles of diaphragmatic crural barrier and esophageal body clearance in patients with gastroesophageal reflux disease]. Zhongguo Yi Xue Ke Xue Yuan Xue Bao. 2002 Jun;24(3):289-93. Chinese. PMID 12905637
- [Background] Ding ZL, Wang ZF, Sun XH, Ke MY. [Therapeutic mechanism of diaphragm training at different periods in patients with gastroesophageal reflux disease]. Zhonghua Yi Xue Za Zhi. 2013 Oct 29;93(40):3215-9. Chinese. PMID 24405544
- [Result] Eherer AJ, Netolitzky F, Hogenauer C, Puschnig G, Hinterleitner TA, Scheidl S, Kraxner W, Krejs GJ, Hoffmann KM. Positive effect of abdominal breathing exercise on gastroesophageal reflux disease: a randomized, controlled study. Am J Gastroenterol. 2012 Mar;107(3):372-8. doi: 10.1038/ajg.2011.420. Epub 2011 Dec 6. PMID 22146488
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials